CLINICAL TRIAL: NCT04892082
Title: Mindful Moment, a Web-based Mindful and Compassionate Parenting Training for Mothers During the Postpartum Period: A Pilot Randomized Controlled Trial
Brief Title: Mindful Moment: Feasibility and Preliminary Efficacy of a Web-based Mindful and Compassionate Parenting Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Daniela Filipa Ventura Fernandes, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MindfulMoment/132588/2017; SFRH/BD/132588/2017 (Other Grant/Funding Number: Foundation for Science and Technology)
Record Dates: First submitted 2021-05-06; First posted 2021-05-19 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Parenting Stress
Keywords: Parenting stress; Mindful Parenting; Compassion; Postpartum period; Mother-infant relationship; eHealth

STUDY DESIGN:
Intervention Model Description: Parallel Assignment - Participants are being randomized to intervention or control groups at a 1:1 ratio
Who Masked: Investigator
Masking Description: Single-blind - the investigator is unaware of the intervention assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Moment (Experimental): Mothers who present parenting stress equal or above 41 score on PSS will receive a web-based intervention to reduce parenting stress (the Mindful Moment program).
  Interventions: Behavioral: Mindful Moment
- Control (Active Comparator): All mothers who present parenting stress will have access to Mindful Moment intervention. The control group only receive the intervention at the end of the intervention group.
  Interventions: Other: Waiting-List Control (WLC)

INTERVENTIONS:
Behavioral: Mindful Moment — The Mindful Moment program is a web-based self-guided cognitive-behavioral intervention to reduce parenting stress, targeting postpartum mothers. It consists of 6 weekly modules, each module targeting a specific thematic content, and providing mothers with both information and specific therapeutic strategies (with a strong focus on the third wave of cognitive-behavioral techniques) to address each thematic content. Modules are sequential.
  Arms: Mindful Moment
Other: Waiting-List Control (WLC) — The control group only receive the intervention at the end of the intervention group.
  Arms: Control

SUMMARY:
Mindful Moment (a web-based mindful and compassionate parenting training) is a self-guided program for postpartum mothers, based on the Mindful Parenting Training developed by Bögels and Restifo (2014) and the Mindful with Your Baby Training (Potharst et al., 2017, 2019). The main goal of this research is to assess the feasibility (e.g., user's adherence, dropout) and acceptability of Mindful Moment and to gather preliminary evidence of its efficacy.

This pilot RCT (Randomized Controlled Trial) will be a two-arm trial. Mothers with a child aged up to 18 months old will be enrolled in the study. A minimum number of 60 mothers will be enrolled in the study. After agreeing to participate in the study, the mothers will be screened for the presence of parenting stress (PSS [Parenting Stress Scale] ≥ 41, Mixão et al., 2007). In case of 41 points score or more, mothers will be asked to complete baseline assessment. Then, mothers who completed baseline assessment will be randomly assigned to one of two conditions: the intervention (Mindful Moment program) or the control condition (Waiting-List control [WLC]). The sample will be recruited online.

The feasibility of Mindful Moment will be evaluated in terms of user's adherence and dropout. Participation in this study will last 16 weeks. The Mindful Moment program will last 8 weeks. Participants in both conditions will be invited via email to complete baseline, post-intervention, and follow-up assessment (8-weeks after post-intervention). Assessments will include self-report questionnaires to assess user's acceptability and satisfaction, several indicators (e.g., parenting stress, depressive and anxiety symptoms, infant's temperament), and mechanisms that may be involved in the treatment response (e.g., mindful parenting, self-compassion).

DETAILED DESCRIPTION:
In the present study, the feasibility (e.g., user's adherence, dropout), acceptability and preliminary efficacy of a web-based intervention to decrease mothers' parenting stress in the postpartum period (the Mindful Moment program) will be tested. The design and content development of the Mindful Moment program was conducted through a formative evaluation process.

Although the birth of a child is a time of great happiness, it is also a period of major adjustment for parents. This period encompasses several demands and reorganizations (e.g., changes in routines, new relationships with partner and family) and psychological and emotional challenges (e.g., ability to regulate the baby's emotional states and one's own internal states). These demands often increase stress levels. It is well-stablished in literature that parenting stress may interfere with sensitive parenting and the ability to form a secure attachment with the child. It is also well-established that the quality of parental care is a major determinant of the child's cognitive, social, and emotional development. Therefore, psychological interventions aimed at helping mothers adjust better to the postpartum period and develop adaptive parenting skills are much needed.

Mindfulness (the capacity to pay nonjudgmental attention to the present moment) and self-compassion (attitude of kindness toward one's suffering and desire to relieve it) skills can be highly beneficial for parents since they are well-known psychological resources that help individuals adaptively cope with stress. Mindful applied to the parenting context can be defined as a more accepting, emotionally attuned, and compassionate way of parenting and it is characterized by parenting practices that promote responsive and sensitive care to the child's needs. Although the scarcity of research during the postpartum period, a few studies have shown that mindful parenting training may reduce mothers' psychopathological symptoms and may promote a more positive mother-infant relationship through the promotion of mindful parenting skills. Likewise, online mindful parenting training seems to be an easily accessible and valuable intervention for mothers with elevated levels of parenting stress including in the postpartum period.

Mindful Moment is a self-guided web-based intervention grounded on CBT (Cognitive-Behavioral Therapy) principles that also includes recent developments in mindfulness and compassion based-therapies, specifically for the postpartum context. This program focuses on the decreasing of parenting stress and the development and enhancement of psychological resources such as mindful parenting and self-compassion.

Mindful Moment is constituted by 6 modules, each module addressing one or two specific thematic contents (1. Mindful parenting and parenting stress; 2. Beginner's mind; 3. Self-compassion and self-care; 4. Reactive vs. responsive parenting; 5. Relationship with others [social support and communication]; 6. Mindful parenting for life). In each module, participants will be provided with both psychoeducational content and therapeutic strategies. Informational material will be given in text format, combined with audio and video.

The main goal of this research is to evaluate Mindful Moment by considering several indicators: 1) Mindful Moment's feasibility in terms of adherence, dropout and the pattern of program usage (e.g., number of completed modules, number of pages accessed in each module); 2) Mindful Moment's acceptability in terms of users' global perceptions of the program; and 3) preliminary evidence of Mindful Moment's efficacy in terms of primary (parenting stress) and secondary outcomes (e.g., mindful parenting; self-compassion; depressive and anxiety symptoms).

The research design of the trial followed the methodological recommendations for the development and evaluation of web-based interventions. A usability test was already conducted through phone-call with 4 mothers who explored the website while verbalizing their experience and opinions (think-aloud sessions). At the end, a brief questionnaire was completed by each participant. The results allowed to identify and implement modifications and the final version of Mindful Moment was achieved, allowing for a pilot RCT efficacy study.

The pilot RCT will be a two-arm trial, conducted with mothers who presented parenting stress (PSS ≥ 41 score). The intervention condition (the Mindful Moment program) will be compared with a control condition (Waiting-List control group). The sample will include mothers who delivered a baby in the postpartum period (up to 18 months postpartum). Mothers are being already recruited online through social media and websites and forums focused on motherhood. The dissemination of the study will also be made in HealthCare Centers, after the approval already obtained from Regional Administration of Health Center (ARS-Center). A minimum number of 30 mothers per condition will be required (N = 60). Accounting for the proportion of mothers who presented moderate or high parenting stress (a total score on PSS of 41 or more) and the 50% of attrition rate over time, an anticipated sample of 600 mothers will be enrolled in the study.

Mothers who demonstrate interest in the study were informed of the study goals, the structure and arms of the research and the researchers' and participants' roles. Mothers who agree to participate in the study gave their informed consent. All ethical requirements for research with humans were guaranteed. Mothers were screened for the presence of parenting stress. In case of lower levels of parenting stress, mothers' participation in the study ended. In case of presenting moderate or high levels of parenting stress (PSS ≥ 41), mothers were randomly assigned (blocked randomization, with allocation concealment) to one of the conditions: the intervention (Mindful Moment program) or the control condition (WLC group).

A researcher (clinical psychologist) will contact mothers in the intervention condition, aiming to explain the program's structure and provide assistance during the course of the study.

Participation in the study will last 16 weeks. The Mindful Moment program will last 8 weeks. Participants in both conditions will be invited via email to complete baseline, post-intervention, and follow-up (8-weeks after post-intervention) assessments. Assessments will include self-report questionnaires to assess user's acceptability and satisfaction, several indicators (e.g., parenting stress, depressive and anxiety symptoms, infant's temperament), and mechanisms that may be involved in the treatment response (e.g., mindful parenting, self-compassion).

ELIGIBILITY:
Inclusion Criteria:

* Having 18 years or more.
* Having a child aged up to 18 months old.
* Being female.
* Being Portuguese.
* Being a resident of Portugal.
* Internet access at home.
* Presence of parenting stress (PSS ≥ 41).

Exclusion Criteria:

* Current diagnosis of serious mental health condition (e.g., schizophrenia, substance abuse, bipolar disorder, and personality disorder).
* Language difficulties that impede comprehension/reading-writing.

All participants will be informed that they will be randomized to one of the study groups and that will only be included if they give informed consent to participate in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 292 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the program for postpartum mothers as measured by adherence and dropout rate | 8 weeks
  Measured through the number of completers and users that dropped out from the web-based intervention before completing it.

SECONDARY OUTCOMES:
Feasibility of the program for postpartum mothers as measured by the pattern of program usage | 8 weeks
  Measured through the number of completed modules, number of pages accessed in each module.
Acceptability of the program for postpartum mothers | 8 weeks
  Measured through specific questions (developed by the researchers) to assess acceptability, based on others web-based intervention studies (e.g., Fonseca et al., 2019; Monteiro et al., 2020). Specifically, participants will be asked questions regarding their intention to use the program (2 items; e.g., "I would use Be a Mom again, if I were to be in a similar situation"), satisfaction with the program (3 items; e.g., "I am satisfied with the help I received at Be a Mom"), usefulness/relevance (5 items; e.g., "Be a Mom has helped me deal with my everyday situations more effectively"), credibility (1 item; "I consider Be a Mom to be a credible program"), and demandingness (1 item; "I feel that participation in Be a Mom was very demanding for me"). Participants answered each question with a Likert-type response scale (from 0 = Not at all applicable to me to 3 = Totally applicable to me). The items of the dimensions comprising more than one item were averaged to compute a dimension score.
Number of mothers with parenting stress using Parenting Stress Scale (PSS) (score ≥ 41) | Baseline
  Measured with Parenting Stress Scale (PSS). The total score ranges between 17 and 85, and higher scores are indicative of higher levels of parenting stress. The authors define 3 levels of parenting stress: a score ranging between 17 and 40 indicates low parenting stress; a score ranging between 41 and 63 indicates moderate parenting stress; and a score ranging between 64 and 85 indicates high parenting stress.
Changes from baseline in the severity of parenting stress | Baseline, 8 weeks, 16 weeks
  Measured with Parenting Stress Scale (PSS). The total score ranges between 17 and 85, and higher scores are indicative of higher levels of parenting stress. The authors define 3 levels of parenting stress: a score ranging between 17 and 40 indicates low parenting stress; a score ranging between 41 and 63 indicates moderate parenting stress; and a score ranging between 64 and 85 indicates high parenting stress.
Changes from baseline in mindful parenting skills | Baseline, 8 weeks, 16 weeks
  Measured with Interpersonal Mindfulness in Parenting Scale for Parents of Infants (IM-P-I). The total score ranges between 28 and 140, and higher scores are indicative of higher levels of mindful parenting.
Changes from baseline in self-criticism and self-compassion | Baseline, 8 weeks, 16 weeks
  Measured with the Self-Compassion Scale - Short Form (SCS-SF). The total score ranges between 1 and 48, and higher scores are indicative of higher levels of self-compassion.
Changes from baseline in mother-infant bonding | Baseline, 8 weeks, 16 weeks
  Measured with the Postpartum Bonding Questionnaire (PBQ). The total score can range between 0 and 60, and higher scores are indicative of a more impaired mother-infant bond.
Changes from baseline in anxiety symptoms | Baseline, 8 weeks, 16 weeks
  Measured with Anxiety Subscale of the Hospital Anxiety and Depression Scale (HADS). The total score for this subscale can range between 0 and 21, and higher scores are indicative of more anxiety symptomatology.
Changes from baseline in depressive symptoms | Baseline, 8 weeks, 16 weeks
  Measured with Edinburgh Postnatal Depression Scale (EPDS). The total score can range between 0 and 30, and higher scores are indicative of more severe depressive symptoms.
Changes from baseline in mindful self-care | Baseline, 8 weeks, 16 weeks
  Measured with Mindful Self-Care Scale - Brief (MSCS-B). The total score range between 24 and 120, and higher scores are indicative of more mindful self-care.
Changes from baseline in dispositional mindfulness | Baseline, 8 weeks, 16 weeks
  Measured with Mindful Attention and Awareness Scale (MAAS). The total score range between 15 and 90, and higher scores are indicative of higher levels of dispositional mindfulness.
Changes from baseline in parenting styles | Baseline, 8 weeks, 16 weeks
  Measured with Infancy Parenting Styles Questionnaire (QDEP-I). The questionnaire contains 5 factors about perceptions and behaviors of parents (Discipline; Parent-led routine; Anxiety; Nurturance; Involvement). Higher scores in the items are indicative of higher scores in the factors.
Changes from baseline in mother's perception of infant temperament | Baseline, 8 weeks, 16 weeks
  Measured with Difficult Infant Temperament Questionnaire. The total score range between 8 and 40, and a higher score is indicative of a more difficult child temperament (perceived by the mother).

CONTACTS AND LOCATIONS:
Overall Officials: Daniela V. Fernandes, MsC, Principal Investigator — Faculty of Psychology and Education Sciences, University of Coimbra
Locations (1):
- Faculty of Psychology and Education Sciences, University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandes DV, Monteiro F, Canavarro MC, Moreira H. A Web-Based, Mindful, and Compassionate Parenting Training for Mothers Experiencing Parenting Stress: Results from a Pilot Randomized Controlled Trial of the Mindful Moment Program. Mindfulness (N Y). 2022;13(12):3091-3108. doi: 10.1007/s12671-022-02016-0. Epub 2022 Nov 10. PMID 36408119